CLINICAL TRIAL: NCT01296737
Title: Validation of Quantitative Ventricular Function Imaging
Brief Title: Validation of Quantitative Ventricular Function Imaging Single Photon Emission Tomography (Spect)Using the D-SPECT Cardiac Camera
Status: Completed | Type: Observational
Sponsor: Spectrum Dynamics (Industry)
Responsible Party: Mathews Fish,MD, PeaceHealth
Other Study IDs: 10-027
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-02

CONDITIONS: Quantitative Validation for Ventricular SPECT Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to validate the use of DSPECT camera for the performance of quantitative spect ventricular function imaging by comparison to a validated procedure performed on standard nuclear cameras.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been referred by their physician to the nuclear medicine department for the quantitative SPECT ventricular function study
* voluntarily participate in the study

Exclusion Criteria:

* voluntarily to the study without being referred to the nuclear medicine department for the quantitative SPECT ventricular function study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients who have been reffered by their physicians to the nuclear medicinew department for the preformance of quantitative SPECT venricular function study and will voluntarily participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear Medicine Department , Sacred Heart Department, Springfield, Oregon, United States